CLINICAL TRIAL: NCT02549326
Title: Vitamin D Intervention in Young Adults With Severe Childhood-onset Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Elisa Holmlund-Suila, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 295/13/03/03/2012
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: Vitamin D
MeSH Terms: conditions — Obesity | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Obese, placebo (Placebo Comparator): Placebo daily for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Obese, vitamin D (Active Comparator): Vitamin D3 50 µg / daily for 12 weeks
  Interventions: Dietary Supplement: vitamin D
- Control, placebo (Placebo Comparator): Placebo daily for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Control, vitamin D (Active Comparator): Vitamin D3 50 µg / daily for 12 weeks
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D
  Other Names: cholecalciferol
  Arms: Control, vitamin D; Obese, vitamin D
Dietary Supplement: Placebo
  Arms: Control, placebo; Obese, placebo

SUMMARY:
Obesity is associated with lower total serum 25-hydroxycholecalciferol (S-25OHD) concentration. However, the impact of obesity on free S-25OHD is inadequately studied. A direct assay for free 25OHD was introduced recently.

The aim of the study was to evaluate differences in vitamin D metabolism between young adults with severe childhood-onset obesity and normal-weight controls. Half of the obese subjects and controls will receive placebo and the other half will receive vitamin D3 50 µg daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* weight-for-height ratio exceeding 60% before the age of 7 years, according to Finnish growth standards and persistence of severe obesity for at least three years in childhood
* referral to the Children's Hospital, Helsinki University Hospital due to severe obesity
* at the age of 7 years lived in the greater Helsinki area

Exclusion Criteria:

* endocrine or genetic disorders underlying obesity (e.g. Prader Willi syndrome, pseudohypoparathyroidism, hypothyroidism, hypercortisolism, diabetes

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
change in S-25OHD | baseline, 6 and 12 weeks
  change in total and free S-25OHD concentrations between obese and controls
baseline S-25OHD | baseline
  differences in total and free S-25OHD between obese and controls

SECONDARY OUTCOMES:
baseline vitamin D-binding protein (DBP) | baseline
  differences in DBP between obese and controls
correlation between S-25OHD and calcium, phosphate, parathyroid hormone (PTH) and osteocalcin | baseline, 6 and 12 weeks
  correlation between S-25OHD (total and free) and calcium, phosphate, PTH and osteocalcin
change in vitamin D-binding protein (DBP) | baseline, 6 and 12 weeks
  change in DBP concentrations between obese and controls

CONTACTS AND LOCATIONS:
Overall Officials: Helena Valta, MD PhD, Study Director — Helsinki University Central Hospital